CLINICAL TRIAL: NCT05117216
Title: Examining the Efficacy of "Technological Parental Monitoring" Approach Versus "Parental Vigilant Care" Approach for Reducing Problematic Internet Usage Among Adolescents
Brief Title: Examining the Efficacy of "Parental Vigilant Care" for Reducing Problematic Internet Usage
Acronym: PVC_PIU_TAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yaron Sela, PhD, Principal Investigator, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PVC_PIU_TAU
Record Dates: First submitted 2021-10-19; First posted 2021-11-11 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Addiction Psychological
Keywords: Problematic Internet Use; Parental Vigilant Care; Parental Training

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Parental Vigilant Care (Experimental): 3 sessions of group parental training
  Interventions: Behavioral: Parental Vigilant Care (Parental training)
- Technological Parental Monitoring (Active Comparator): The installation of filtering devices on adolescents' mobile phones and setting them for reducing time use and prohibiting inappropriate content
  Interventions: Behavioral: Technological Parental Monitoring
- PVC + TPM (Active Comparator): combining both group parental training and installation of filtering devices
  Interventions: Behavioral: Parental Vigilant Care (Parental training); Behavioral: Technological Parental Monitoring
- Control (No Intervention): Control group that did not receive any intervention

INTERVENTIONS:
Behavioral: Parental Vigilant Care (Parental training)
  Arms: PVC + TPM; Parental Vigilant Care
Behavioral: Technological Parental Monitoring
  Arms: PVC + TPM; Technological Parental Monitoring

SUMMARY:
Problematic Internet Use (PIU) and Unsafe Internet Use (UIU) are the two main potential negative consequences of children's online activities. Parents have a vital role in reducing these consequences and shaping a safe digital environment. Parental Vigilant Care (PVC) is a systematic approach that integrates active and restrictive mediation practices, in which parents regulate their involvement according to the alarm signs the parents detect.

This study is a randomized controlled trial designed to assess the efficacy of the PVC parent training. Families were randomly assigned to either (1) PVC group (2) Technological Parental Monitoring group (3) combining both group parental training and installation of filtering devices (PVC + TPM) or (4) Control group.

DETAILED DESCRIPTION:
BACKGROUND: One of the most disturbing phenomena regarding the digital age is Problematic Internet Use (PIU) among adolescents (12-16). PIU is defined as a functioning impairment due to: (1) internet excessive use that may lead to the neglect of developmental tasks, or (2) unsafe use which includes viewing inappropriate content, abusive encounters, or commercial exploitation. Clinical and research experience shows that parental involvement plays a critical role in reducing risk behaviors among adolescents in various domains. Despite the ample literature regarding parental involvement, few studies have evaluated the efficacy of parental involvement on adolescents' PIU in reducing functional impairment and designing a safe digital environment. One of the most investigated theoretical approaches in this field is Parental Monitoring (PM). PM is defined as a set of parental practices that aim to monitor and supervise adolescent activities. Despite evidence that PM is effective in reducing risk behaviors among adolescents, PM also has some drawbacks. Studies have demonstrated that it may be perceived as rigid parental control, thereby damaging internalization of parental presence, and potentially sabotaging adolescents' growing independence and autonomy. In the digital world, rigid PM can be defined as using filtering and surveillance applications that enable parents to closely monitor and enforce strict rules regarding their child's internet use. This approach is defined as in the current study as "Technological Parental Monitoring" (TPM). On the other hand, "Parental Vigilant Care" (PVC), is theoretically conceptualized as an alternative parental involvement approach that addresses the weaknesses of PM. By implementing PVC principles, parents develop a positive and non-judgmental dialogue with their children regarding domains the participants are concerned about. Additionally, parents determine their level of active involvement in a flexible manner, specific to the risks presented by their children. By executing decisive and consistent parental involvement, parents strengthen their presence in their children's digital world, therefore, reducing PIU by internalization of safe digital behavior.

OBJECTIVES: The current study aims to examine the efficacy of using digital parental control, according to TPM approach, in comparison with flexible integration of positive parental presence with setting boundaries, according to PVC approach. These approaches will be compared in light of the following outcomes: (1) increasing effective parental involvement in PIU of their adolescent children, (2) reducing PIU and improving adolescent's functioning, and (3) internalizing parental values regarding safe digital activities by children, in order to maintain a parental presence over time.

METHOD: To examine these objectives, a randomized controlled trial was conducted.

Sample size calculation: To assess sample size, the investigators used G-Power software, assuming type 1 error of 5%, power 80%, and analysis of variance, repeated measures with three measurement points, a moderate effect size of time X group interaction (µ2 = .15). The minimum sample size required to meet these assumptions was 134 participants. The final sample consisted of 157 adolescents, in addition to their parents (one parent for each adolescent), yielding a total sample size of 314 participants.

Two-hundred and 297 parents and their children (12-16 y/o) were randomly assigned to four groups: (1) Group parental training according to PVC approach; (2) installation of filtering devices on adolescents' mobile phones and setting them for reducing time use and prohibiting inappropriate content (TPM); (3) combining both group parental training and installation of filtering devices (PVC + TPM) and (4) control group that did not receive any intervention.

Three types of measures were used: (A) Self-reported questionnaires completed by parents: Parental Helplessness for Internet Supervision, Internet Parental Styles, Norms for Unsafe Internet Behaviour, Parental Knowledge of the child's online activities, Family Environment and Adolescent's Functioning (B) Self-reported questionnaires completed by adolescent: Problematic Internet Use and unsafe internet behavior (C) Cellular internet usage retrieved directly from adolescents' mobile devices including total time online, as well as time by specific contents (video games, pornography, gambling, YouTube and social networking sites). The self-report questionnaires were gathered at three time points - before intervention (T1), immediately after termination of intervention (T2) and after 8 weeks follow-up (T3). The online activities data were gathered continuously for 12 weeks (a baseline week, 3 weeks of intervention and 8 weeks of follow-up).

Data Analysis:

Data were analyzed using SPSS version 25. First, descriptive statistics were produced using means and standard deviations for all variables. Group comparisons on demographic variables were conducted using chi-square tests for categorical variables and t- tests for continuous variables. Intervention effects were examined using intent-to-treat analyses. The groups were compared with self-reported measures using repeated measures Analysis of Covariance, examining interaction effect between time (within-subject) and group (between-subject). In these analyses, the expectation to benefit from treatment was controlled. Post-hoc corrections were used for to further examine the significant two-way interactions, and depicted the effect sizes using Cohen's d's both between baseline (T0) and post-intervention (T1), and also between post-intervention (T1) and follow-up (T2). Time of online activity was analyzed using Multi-Level Modeling (MLM) since average daily time online per-week (12 weeks) was nested in the child's group (PVC vs. Control). In addition, to examine the persistence of improvement achieved during intervention, change in average time online between intervention period (3 weeks) and the follow-up period (8 weeks) was tested.

ELIGIBILITY:
Inclusion Criteria:

* Functioning deterioration of the child (age 12-16) due to online activity in the past 6 months in at least one of the following domains: school, social relationships, participation in family activities, sleeping patterns, and mood (according to parents' self-report).
* The child owns a mobile phone.

Exclusion Criteria:

* A psychiatric diagnosis of the child
* A significant personal crisis in the previous 12 months (e.g., divorce, loss of a significant person)
* A parental control application is installed on their children's mobile phones.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Internet use (hours/day) by Adolescence | Reducing time online, through study completion, an average of 12 weeks
  Time online using mobile

SECONDARY OUTCOMES:
Parental Helplessness for Internet Supervision | Improving parental helplessness, through study completion, an average of 12 weeks
  Self-reported scale: 1-Lowest Parental Helplessness, to 7-Most severe Parental Helplessness
Adolescent's Functioning Impairment | Improving adolescent's functioning, through study completion, an average of 12 weeks
  Self-reported scale: 1-Mild Functioning Impairment , to 7-Most severe Functioning Impairment
Family Environment | Improving family environment, through study completion, an average of 12 weeks
  Self-reported scale: 1- Poor Family Environment , to 7-Extremely Positive Family Environment

CONTACTS AND LOCATIONS:
Overall Officials: Meir Lahav, Prof., Study Chair — Tel Aviv University

IPD SHARING:
Plan to Share IPD: No